CLINICAL TRIAL: NCT00421603
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Mixed Amphetamine Salts (Adderall-XR) and Topiramate for the Treatment of Cocaine Dependence
Brief Title: A Placebo-Controlled Study of Mixed Amphetamine Salts and Topiramate for the Treatment of Cocaine Dependence
Acronym: TACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #5368; R01DA022217 (NIH)
Record Dates: First submitted 2007-01-10; First posted 2007-01-12 (Estimated); Results first posted 2013-02-28 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; Adderall; Topiramate; ADHD
MeSH Terms: conditions — Cocaine-Related Disorders; Attention Deficit Disorder with Hyperactivity | interventions — SLI381; Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adderall-XR and Topiramate (Active Comparator): Adderall-XR (60 mg/day) and Topiramate (300mg/day)
  Interventions: Drug: Adderall-XR and Topiramate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adderall-XR and Topiramate — Adderall-XR 60mg/day and Topiramate 300mg/day
  Arms: Adderall-XR and Topiramate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The proposed protocol is a double-blind, placebo-controlled outpatient study of the safety and efficacy of Adderall-XR (ER-MAS) and topiramate in the treatment of cocaine dependence. Since both of these medications have independently shown promise in helping with cocaine abuse we are proposing that together they may be even more successful in the treatment of cocaine abuse. We plan to enroll 120 subjects in a 14-week trial. The primary objective of the study is to determine the efficacy of ER-MAS and topiramate in promoting cocaine abstinence among cocaine-dependent patients. This study includes free treatment for cocaine dependence that includes medication.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the efficacy of ER-MAS and topiramate in promoting cocaine abstinence among cocaine-dependent patients.

Primary Hypothesis: The proportion of participants achieving sustained cocaine abstinence (via urine toxicology) for three consecutive weeks during the study will be significantly greater for the combined pharmacotherapies group compared to the placebo group.

Hypothesis 2: The proportion of urine samples negative for cocaine metabolites will be greater in the combined pharmacotherapies group compared to the placebo group.

Hypothesis 3: The pattern of cocaine use (amount of cocaine used per day in dollars and the number of using days per week), as measured by the time-line follow-back method, will show a greater reduction in use for the combined pharmacotherapies group compared to the placebo group.

Specific Aim 2: To determine the effect of ER-MAS and topiramate on cocaine craving among cocaine-dependent patients.

Hypothesis 4: Cocaine craving symptoms will be reduced to a greater degree in the combined pharmacotherapies group compared to the placebo group.

Specific Aim 3: To explore a set of related secondary outcomes (treatment retention, global functioning, HIV risk behavior) as well as moderators and mediators potentially reflective of mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-60 who meet DSM-IV criteria for current cocaine dependence (DSM-IV-TR).
2. Used cocaine at least four days in the past month, with at least weekly cocaine use.
3. Must have a Body Mass Index (BMI) > 18 kg/m2
4. Alcohol Breathalyzer (BraC) at consent of < 0.04%
5. Individuals must be capable of giving informed consent and capable of complying with study procedures.
6. Women of child bearing age will be included in the study provided that they are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, blood pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study medication. If a woman becomes pregnant, the study medication will be discontinued.

Exclusion Criteria:

1. Meets DSM-IV-TR criteria for bipolar disorder, Schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse
2. Individuals with any current Axis I psychiatric disorder as defined by DSM-IV-TR supported by the SCID-I/P that in the investigator's judgment are unstable or would be disrupted by study medication or are likely to require pharmacotherapy during the study period.
3. Individuals with current major depressive disorder.
4. Individuals physiologically dependent on any other drugs (excluding nicotine or cannabis) which require medical intervention.
5. Individuals with current psycho stimulant abuse or dependence.
6. Individuals with current suicidal risk.
7. Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms.
8. Unstable physical disorders which might make participation hazardous such as uncontrolled hypertension (SBP > 150, DBP> 90, or HR > 100 when sitting quietly), acute hepatitis (patients with chronic mildly elevated transaminases < 3x upper limit of normal are acceptable), or uncontrolled diabetes.
9. Individuals with a history of seizures
10. History of allergic reaction to candidate medication (amphetamine and/or ER-MAS or topiramate).
11. Women who are pregnant or nursing.
12. Use of carbonic anhydrase inhibitors*
13. History of glaucoma, kidney stones*
14. History of failure to respond to a previous Adequate trial of either candidate medication for Cocaine dependence
15. Currently being prescribed psychotropic medication by another physician (other than sleep medication)
16. Individuals who are legally mandated (e.g., to avoid incarceration, monetary or other penalties, etc.) to participate in substance abuse treatment program -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2007-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

REFERENCES:
- See also: Substance Treatment and Research Service of Columbia University — http://www.stars.columbia.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by local advertising (internet, print, radio, television, and subway) or by clinical referrals in the New York City metropolitan area between January 2007 and February 2010.
Pre-assignment Details: Prior to group assignment patients participated in a one week placebo lead-in.
Groups:
- Adderall-XR and Topiramate: Adderall-XR doses were titrated over two weeks to a maximum dose of 60 mg daily and topiramate doses were titrated over six weeks to a maximum dose of 150 mg twice daily.
- Placebo: Placebo daily dose
Period: Overall Study
Arm/Group | Adderall-XR and Topiramate | Placebo
Started | 39 | 42
Completed | 28 (Completed all 14 week sof trial) | 30 (Completed all 14 week sof trial)
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adderall-XR and Topiramate | Placebo | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 42 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (8.2) | 42.4 (8.9) | 42.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 33 | 37 | 70
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Three Weeks of Continuous Cocaine Abstinence as Measured by Urine Toxicology and Self Report Based on Time Line Follow Back
Description: Cocaine use was assessed by using urine toxicology confirmed self-report. Self-reported cocaine use data was collected for each day of the study period by the Time Line Follow Back. Urine samples were collected three times per week. A week was considered abstinence if no cocaine use was self reported during that week and if all urine samples collected that week were negative for cocaine. If a patient achieved three continuous weeks of abstinence based on this criteria they were considered cocaine abstinent in terms of this outcome measure.
Time Frame: 3 weeks of abstinence during 14 weeks of trial or for length of participation
Measure: Number; unit: participants
Arm/Group | Adderall-XR and Topiramate | Placebo
Number analyzed (Participants) | 39 | 42
participants | 13 | 7
Statistical Analysis 1: Comparison: Adderall-XR and Topiramate vs Placebo; The dichotomous primary outcome was analyzed using logistic regression with independent predictors: treatment (MAS-ER and topiramate vs. placebo) and adjusted for baseline severity of cocaine use (total number of cocaine use days in the 28 days prior to randomization); Test type: Non-Inferiority or Equivalence — All analyses were conducted on the intent-to-treat sample of all randomized patients. All statistical tests were 2-tailed and employed at a significance level of 5%, unless otherwise stated. The original sample size of 120 patients was chosen to ensure sufficient power (at least 80%) of a two-sided test with level of significance α=0.05 for detecting difference between the two experimental treatments with respect to the percentage of subjects who achieve continuous 3-weeks abstinence; p = .05, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: during 14 weeks of trial or length of participants participation
Arm/Group | Adderall-XR and Topiramate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/39 | 1/42
Other Adverse Events (participants affected / at risk) | 33/39 | 21/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adderall-XR and Topiramate (N=39) | Placebo (N=42)
substance-induced mood syndrome (Psychiatric disorders) | 1 (1) | 0 (0) — One participant in the MAS-ER and topiramate group developed a substance-induced mood syndrome and required hospitalization.
residential drug treatment (Psychiatric disorders) | 0 (0) | 1 (1) — The other participant in the placebo group voluntarily discontinued study participation during the final week of the trial and entered a residential substance abuse treatment center.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adderall-XR and Topiramate (N=39) | Placebo (N=42)
Insomnia (Psychiatric disorders) | 16 (16) | 7 (7)
Increased/decreased appetite (Metabolism and nutrition disorders) | 17 (17) | 4 (4)
Fatigue (General disorders) | 11 (11) | 6 (6)
GI upset (Gastrointestinal disorders) | 11 (11) | 5 (5)
Headache (General disorders) | 11 (11) | 5 (5)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (4)
Dizziness (General disorders) | 10 (10) | 4 (4)
Anxiety (Psychiatric disorders) | 9 (9) | 1 (1)
Paresthesia (Nervous system disorders) | 9 (9) | 1 (1)
Irritable (General disorders) | 8 (8) | 2 (2)

LIMITATIONS AND CAVEATS:
The two-arm placebo controlled design does not allow us to address whether both medications are necessary for efficacy. Potential limited treatment masking that occurred when giving two medications with distinctive adverse effect profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No